CLINICAL TRIAL: NCT05562414
Title: Transient and Immediate Motor Effects of Exercise in Progressive Multiple Sclerosis: A Pilot Study.
Brief Title: Transient and Immediate Motor Effects of Exercise in Progressive Multiple Sclerosis
Acronym: TIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, Jens Bansi, Dr. Jens Bansi, Head of Research and Development, Klinik Valens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIME
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis, Chronic Progressive; High-Intensity Interval Training; Motor Symptoms
Keywords: Multiple Sclerosis, Chronic Progressive; Physical Conditioning, Human; Paraparesis; Gait; Dexterity
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Motor Activity; Paraparesis

STUDY DESIGN:
Intervention Model Description: Single-centre Randomized Controlled Trial (RCT)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of the principal investigator and research assistant towards group allocation is ensured by a unique subject identification code given to each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity Interval Training (HIIT) (Experimental): Participants will complete one heart-rate-controlled HIIT bout within their 3-week inpatient stay.
  Interventions: Behavioral: HIIT
- Moderate Continuous Training (MCT) (Active Comparator): MCT represents the standard treatment at Valens rehabilitation clinic. Participants will complete one heart-rate-controlled MCT bout within their 3-week inpatient stay.
  Interventions: Behavioral: MCT

INTERVENTIONS:
Behavioral: HIIT — Exercise intensity will be regulated and heart rate controlled based on the age-predicted heart rate (HRmax), as calculated by the formula 220 minus age in years.
  Participants will perform six high-intensity intervals (95% HRmax) at high pedalling rates of 80-100 rounds per minute (rpm) for 60-90 seconds each. Intervals are interspersed by active breaks of unloaded pedalling (20 watts, 60-80rpm) aimed to return to 60% HRmax (approximately 1.5-2 min). The duration of the HIIT bout is approximately 21 minutes.
  Arms: High-intensity Interval Training (HIIT)
Behavioral: MCT — Exercise intensity will be regulated and heart rate controlled based on the age-predicted heart rate (HRmax), as calculated by the formula 220 minus age in years.
  Participants will continuously train at 60% HRmax and pedal at 60-80 rounds per minute. The duration of the MCT bout is 26 minutes.
  Arms: Moderate Continuous Training (MCT)

SUMMARY:
Endurance training is a cornerstone of rehabilitation in Multiple Sclerosis (MS) due to its beneficial effects on multiple MS-related symptoms, such as health-related quality of life, aerobic capacity (VO2peak), functional mobility, gait, depressive symptoms, and fatigue.

Persons with progressive phenotypes of MS, namely primary progressive MS (PPMS) and secondary progressive (SPMS), represent a minor proportion of the total MS population, thus having been underrepresented in previous studies. The generalizability of existing evidence may be compromised by differences in symptom expression between MS phenotypes, with a dominance of motor symptoms (i.e., paraspasticity and/or paraparesis) in PPMS and SPMS.

Adding up to this, clinical experiences of neurologists and sports scientists reveal that the effects of endurance exercise are characterized by a distinct time course, firstly inducing a minor and transient deterioration of motor symptoms that is followed by motor symptom alleviation beyond baseline level. This phenomenon was mainly related to the performance of High-Intensity Interval training (HIIT), but not to moderate-intensity continuous training (MCT).

Therefore, this pilot study aims to systematically investigate the time course of acute motor effects on spasticity, functional mobility, gait, and dexterity in persons with PPMS and SPMS following two different endurance training protocols, that are HIIT and MCT.

ELIGIBILITY:
Inclusion Criteria:

* adult age (≥ 18 years)
* definite MS diagnosis according the 2017 revised McDonald criteria
* PPMS/SPMS phenotype according to the 2013 revised Lublin criteria
* Expanded Disability Status Scale (EDSS) score ≤ 6.0
* Informed Consent as documented by signature of participants and PI

Exclusion Criteria:

* severe lower extremity spasticity or severe concomitant disease states (i.e., orthopaedic, cardiovascular, metabolic, psychiatric (e.g., substance abuse), other neurological, other serious medical conditions) impairing the ability to participate
* inability to follow study procedures (e.g., due to language barriers)
* suspected non-compliance
* previous enrolment into the current study
* enrolment of the investigator, his/her family members, employees, and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Functional mobility | Change from baseline to directly after, 1-hour after, 3-hours after, and 5-hours after the exercise bout
  Functional mobility is assessed by the Timed-Up-and-Go Test (TUG). For the TUG, participants are asked to get up from a chair, walk a 3 metres distance, perform a 180° turn, return to the chair, and sit down again as fast as possible. Assessment takes place on a single day, before (T0), 5 minutes after (T1), 60 minutes after (T2), 180 minutes after (T3), 300 minutes (T4) after HIIT/MCT cycling bout.

SECONDARY OUTCOMES:
Spasticity (objective) | Change from baseline to directly after, 1-hour after, 3-hours after, and 5-hours after the exercise bout
  Spasticity of the hip flexors, knee flexors, foot dorsiflexors and respective extensors will be evaluated using the Modified Ashworth Scale (MAS). The participant is placed on a bench in supine position. The outcome assessor performs a passive stretch on the respective muscle group and scores the muscle tone as normal or increased on a 6-category ordinal scale (0, 1, 1+, 2, 3, 4). Assessment takes place on a single day, before (T0), 5 minutes after (T1), 60 minutes after (T2), 180 minutes after (T3), 300 minutes (T4) after HIIT/MCT cycling bout.
Spasticity (subjective) | Change from baseline to directly after, 1-hour after, 3-hours after, and 5-hours after the exercise bout
  Participants rate the extent of perceived spasticity on a Numeric Rating Scale for Spasticity (NRS-S), ranging from 0 ("no spasticity") to 10 ("worst possible spasticity"). Assessment takes place on a single day, before (T0), 5 minutes after (T1), 60 minutes after (T2), 180 minutes after (T3), 300 minutes (T4) after HIIT/MCT cycling bout.
Gait pattern | Change from baseline to directly after, 1-hour after, 3-hours after and 5-hours after the exercise bout
  Spatiotemporal features of the gait pattern analysis are captured by the instrumented treadmill C-Mill for a duration of two minutes. Assessment takes place on a single day, before (T0), 5 minutes after (T1), 60 minutes after (T2), 180 minutes after (T3), 300 minutes (T4) after HIIT/MCT cycling bout.
Dexterity | Change from baseline to directly after, 1-hour after, 3-hours after, and 5-hours after the exercise bout
  Dexterity is assessed by the Virtual Peg Insertion Test (VPIT). The VPIT is a virtual instrumented 3D object manipulation (pick-and-place) task. In seated position, participants are asked to transport virtual pegs into virtual holes as fast as possible. Participants perform four trials with their dominant hand. Spatiotemporal movement trajectories are recorded. Assessment takes place on a single day, before (T0), 5 minutes after (T1), 60 minutes after (T2), 180 minutes after (T3), 300 minutes (T4) after HIIT/MCT cycling bout.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gonzenbach, MD, Principal Investigator — Kliniken Valens
Locations (1):
- Klinik Valens, Valens rehabilitation clinic, Valens, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heine M, van de Port I, Rietberg MB, van Wegen EE, Kwakkel G. Exercise therapy for fatigue in multiple sclerosis. Cochrane Database Syst Rev. 2015 Sep 11;2015(9):CD009956. doi: 10.1002/14651858.CD009956.pub2. PMID 26358158
- [Background] Ensari I, Motl RW, Pilutti LA. Exercise training improves depressive symptoms in people with multiple sclerosis: results of a meta-analysis. J Psychosom Res. 2014 Jun;76(6):465-71. doi: 10.1016/j.jpsychores.2014.03.014. Epub 2014 Mar 31. PMID 24840141
- [Background] Latimer-Cheung AE, Pilutti LA, Hicks AL, Martin Ginis KA, Fenuta AM, MacKibbon KA, Motl RW. Effects of exercise training on fitness, mobility, fatigue, and health-related quality of life among adults with multiple sclerosis: a systematic review to inform guideline development. Arch Phys Med Rehabil. 2013 Sep;94(9):1800-1828.e3. doi: 10.1016/j.apmr.2013.04.020. Epub 2013 May 10. PMID 23669008
- [Background] Taul-Madsen L, Connolly L, Dennett R, Freeman J, Dalgas U, Hvid LG. Is Aerobic or Resistance Training the Most Effective Exercise Modality for Improving Lower Extremity Physical Function and Perceived Fatigue in People With Multiple Sclerosis? A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2021 Oct;102(10):2032-2048. doi: 10.1016/j.apmr.2021.03.026. Epub 2021 Apr 24. PMID 33901439
- [Background] Ward M, Goldman MD. Epidemiology and Pathophysiology of Multiple Sclerosis. Continuum (Minneap Minn). 2022 Aug 1;28(4):988-1005. doi: 10.1212/CON.0000000000001136. PMID 35938654
- [Background] Bansi J, Koliamitra C, Bloch W, Joisten N, Schenk A, Watson M, Kool J, Langdon D, Dalgas U, Kesselring J, Zimmer P. Persons with secondary progressive and relapsing remitting multiple sclerosis reveal different responses of tryptophan metabolism to acute endurance exercise and training. J Neuroimmunol. 2018 Jan 15;314:101-105. doi: 10.1016/j.jneuroim.2017.12.001. Epub 2017 Dec 6. PMID 29224960